CLINICAL TRIAL: NCT06532708
Title: Prospective Study of Opioid Prescribing Practices in Laparoscopic Gynecologic Surgery
Brief Title: Opioid Prescribing Practices in Laparoscopic Gynecologic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-09978-FB
Record Dates: First submitted 2024-07-15; First posted 2024-08-01 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Opioid Use; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 5 Doses (Experimental): Participants will receive 5 doses of prescription opioids following surgery.
  Interventions: Other: 5x Oxycodone Oral Tablets
- 16 Doses (Active Comparator): Participants will receive 16 doses of prescription opioids following surgery.
  Interventions: Other: 16x Oxycodone Oral Tablets

INTERVENTIONS:
Other: 5x Oxycodone Oral Tablets — Participants will be prescribed 5 doses of 5mg tablets of oxycodone for postoperative pain relief.
  Arms: 5 Doses
Other: 16x Oxycodone Oral Tablets — Participants will be prescribed 16 doses of 5mg tablets of oxycodone for postoperative pain relief.
  Arms: 16 Doses

SUMMARY:
The purpose of this study is to compare opioid prescribing practices by either routine provider prescribing practices, or with the use of a calculator, i.e., the Opioid Calculator, published by the University of Michigan (www.opioidcalculator.org), with the intent of decreasing the number of pills.

DETAILED DESCRIPTION:
The intent of this study is to validate the use of the Opioid Calculator, published at University of Michigan (www.opioidcalculator.org), which takes several variables into account, including age, risk factors (history of depression, alcohol abuse, others) to determine in a more scientific way the number of pills sufficient to prescribe. The sample size was determined by the number of routine post-op laparoscopic patients seen in our practice. The estimated necessary sample size is 6 participants per group (12 total). Patients will be randomized using 3 block groups of size 4 each. Patients will be approached at in clinic at the time they are consenting to laparoscopic hysterectomy and will be counseled about postoperative pain medication management. Randomization to either standard practice or calculator will be performed using computer-generated, permuted blocks of 4 participants. Sealed randomization envelopes will be opened for each subject on the day of surgery, after anesthesia is initiated. The study will be singled-blinded to the participant. Patients will be contacted on day 2 and day 7 to inquire where they are on the Visual Analog Scale (VAS) and how many pills they have taken. Two weeks after surgery patients will be seen in office for VAS and requested to bring unused pills for accounting purposes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 80
* Undergoing planned laparoscopic hysterectomy as a day surgery procedure

Exclusion Criteria:

* Women aged 18 to 80
* Undergoing a non-laparoscopic unplanned surgical procedure
* Patients with a history of opioid use disorder or current opioid use disorder

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are biologically female
Enrollment: 12 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of pills used | Within 1 week following surgery
  All participants will be contacted on postoperative days 2 and 7 to inquire how many pills they have taken

SECONDARY OUTCOMES:
Postoperative pain | Within 2 weeks following surgery
  All participants will be contacted on postoperative days 2 and 7, and at their two-week follow-up visit to inquire where their pain level is on the Visual Analog Scale (VAS). This scale ranges from 0 to 10, with 0 indicating no pain and 10 indicating worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Straubhar AM, Stroup C, de Bear O, Dalton L, Rolston A, McCool K, Reynolds RK, McLean K, Siedel JH, Uppal S. Provider compliance with a tailored opioid prescribing calculator in gynecologic surgery. Gynecol Oncol. 2023 Mar;170:229-233. doi: 10.1016/j.ygyno.2023.01.018. Epub 2023 Jan 28. PMID 36716511
- [Background] Wong M, Vogell A, Wright K, Isaacson K, Loring M, Morris S. Opioid use after laparoscopic hysterectomy: prescriptions, patient use, and a predictive calculator. Am J Obstet Gynecol. 2019 Mar;220(3):259.e1-259.e11. doi: 10.1016/j.ajog.2018.10.022. Epub 2018 Oct 25. PMID 30837064

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT06532708/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT06532708/ICF_001.pdf